CLINICAL TRIAL: NCT01280890
Title: Person-centred Care and Dementia Care Mapping Among Nursing Home Patients - a 10 Months Randomised Controlled Intervention Study
Brief Title: Person- Centred Care Among Nursing Home Patients With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Centre for Ageing and Health (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PCCNor; 196326/V50 (Other Grant/Funding Number: The Research Counsil of Norway)
Record Dates: First submitted 2011-01-18; First posted 2011-01-21 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Dementia; Agitation
Keywords: Dementia; Nursing home; Person-centred Care; Staff training
MeSH Terms: conditions — Dementia; Psychomotor Agitation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Staff training using VIPS framework (Experimental): The staff will be trained to give person-centred care using the VIPS framework
  Interventions: Behavioral: Staff training using VIPS
- Staff training using DCM (Experimental): Staff will be supervised in how to give person-centred care using Dementia Care Mapping
  Interventions: Behavioral: Staff training using DCM
- Control group (Placebo Comparator): Traditional lectures using films will be given to care staff
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Staff training using VIPS — Staff training using the VIPS framework
  Other Names: Person-centred care; Dementia care
  Arms: Staff training using VIPS framework
Behavioral: Staff training using DCM — The staff will be supervised using Dementia Care Mapping
  Other Names: Person-centred Care; dementia Care
  Arms: Staff training using DCM
Behavioral: Control group — Filmed traditional Lectures will be given to care staff
  Other Names: Staff training
  Arms: Control group

SUMMARY:
Dementia is a common and devastating disease in the elderly. No cure exist and there is an increasing need for care. To improve knowledge on how to provide better care for the patients with dementia in nursing homes, the investigators will carry out a controlled trial using two forms of education and developmental interventions towards the nursing home care staff: a structured framework (VIPS) and dementia care mapping (DCM)to develop person-centred care in a 10 months randomised controlled study. In accordance with the knowledge found in the literature the investigators hypothesize that both VIPS framework and DCM will be more effective than a traditional educational program about dementia provided to the staff in nursing homes. The positive effects will be seen as reduced agitation in patients, less use of psychotropic drugs and improved quality of life. Using VIPS framework and DCM will also have a better effect on staffs' well-being than traditional education in dementia. The aim of the study is to confirm or reject these hypotheses.

DETAILED DESCRIPTION:
This is a controlled intervention trial with three groups of staff recruited from 15 nursing homes in the city of Oslo. The intervention will be carried out over 10 months. Randomization will be done at institutional level. Before randomization all patients in the participating nursing homes should be screened for dementia. This will be done by interviewing the registered nurses in the nursing homes using the Clinical dementia rating scale (CDR), Neuropsychiatric inventory (NPI-Q), Cornell scale for depression in dementia (CSDD). In addition information from the records will be used. Diagnosis of dementia will be made according to ICD-10 criteria, using a diagnostic algorithm that is evaluated in an ongoing nursing home study.

The nursing homes will be randomized in tree groups. Group A - Applying the VIPS- framework to develop Person Centred Care (PCC) and milieu therapy. The staff will be introduced to the model for applying the VIPS-framework to promote PCC in the daily care. A manual including films with information and examples will be distributed to all staff. Two auxiliary nurses are appointed as resource persons (RP) from each ward and one registered nurse (RN) from each nursing home will be trained as coach. The RPs and the leading registered nurse (RN) will plan and lead weekly consensus meetings with the staff in the ward using the VIPS-framework in discussions of concrete care situations. The researches will receive monthly written standard reports on attendance and contents of the consensus meetings from the RPs and can be contacted for support when necessary.

Group B - using Dementia Care Mapping (DCM) developing Person Centred Care and milieu therapy All staff and leaders in the nursing home will be introduced to the DCM- process in a presentation of the method and person centred care as a value base for DCM. A group of 3-5 staff members from each nursing home will be trained as DCM basic users. Dementia Care Mappings (4-6 hours) will be made in each unit in the nursing homes and feed-back (1, 5 hours) will be given to the staff within a week after the mapping. Based on the findings and the reflections in the feed-back session, action plans on how to develop care to selected patients and/or to the group of patients, will be created in the units. The project leader will be responsible for the introduction, mapping and feed-back sessions and give the necessary supervision to create action plans. The leaders and staff in the nursing home units will be responsible for the implementation of the changes to develop practice.The DCM-process will be repeated after 6-8 months

Group C (control group) - traditional education Lectures made as 5 DVD films lasting for 30 minutes, will be given to the nursing home staff on three themes: types of dementia, legal aspects of use of restraints and challenging behavior

The staff in group A and B will receive the same lectures as the staff in the control group.

Effect will be measured on patient and staff level, and measurements will be done at baseline and after 10 months of intervention. Data will be collected by research assistants, who will not take part in the three different intervention programs and not be employed by the nursing homes that are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Persons with dementia living in nursing homes
* A score of 1,2 or 3 on the Clinical Dementia Rating Scale (CDR)
* The nursing staff in the wards where the patients are

Exclusion Criteria:

* Result from the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 624 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in agitation at 10 months from baseline using Brief Agitation Rating Scale | After 10 months
  Brief Agitation Rating Scale (BARS)will be used to measure change in agitation from basline to end of intervention after 10 months

SECONDARY OUTCOMES:
Neuropsychiatric Inventory (NPI-Q) | After 10 months
Cornell scale for depression in dementia | After 10 months
Quality of life in Alzheimer's Disease (QUALID) | After 10 months
Use of psychotropic drugs | After 10 months
  collected from the patients' records
Clinical Dementia Rating Scale (CDR) | After 10 months
Lawton maintenance scale | After 10 months
  Measures function in activities of daily living
Person-centred Care Assessment Tool (P-CAT) | after 10 months
QPSNordic | After 10 months
  A scale developed to measure psychological and social factors in working life
Stress of Conscience Questionaire (SCQ) | After10 months
  Assessing stressful situations experienced by staff and the degree to which they trouble the conscience

CONTACTS AND LOCATIONS:
Overall Officials: Knut Engedal, Dr.med, Principal Investigator — Norwegian Centre for Ageing and Health